CLINICAL TRIAL: NCT06803888
Title: Efficacy and Safety of Bariatric Surgery, Semaglutide Once Weekly, and Tirzepatide Once Weekly in Patients With Obesity
Brief Title: Bariatric Surgery vs. Semaglutide vs. Tirzepatide
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ali Aminian (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ali Aminian, Director of the Bariatric and Metabolic Institute, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-915
Record Dates: First submitted 2025-01-14; First posted 2025-01-31 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Obesity and Obesity-related Medical Conditions
Keywords: Bariatric Surgery; Tirzepatide; Semaglutide; Obesity; GLP-1 Receptor Agonist; Mounjaro; Wegovy; Zepbound; Ozempic; Sleeve Gastrectomy; Roux-en-Y gastric bypass
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery; Gastric Bypass; semaglutide; Tirzepatide

STUDY DESIGN:
Intervention Model Description: This is a randomized non-blinded controlled efficacy/safety study with 3 parallel groups who will either receive bariatric surgery (RYGB or SG), semaglutide, or tirzepatide. The study has 2 phases: the first 12 months for the assessment of the primary endpoint, and the second 12 months as the extension phase of the study to mimic the real-life setting. Findings at the end of each phase will be separately reported.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bariatric Surgery (Active Comparator): Roux-en-Y Gastric Bypass (RYGB) and Sleeve Gastrectomy (SG)
  Interventions: Procedure: Bariatric Surgery
- Semaglutide (Active Comparator): Semaglutide, which is an incretin-based medication that has been approved for the treatment of obesity, will be used for this arm.
  Interventions: Drug: Semaglutide
- Tirzepatide (Active Comparator): Tirzepatide, which is an incretin-based medication that has been approved for the treatment of obesity, will be used for this arm.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Procedure: Bariatric Surgery — Patients receive either RYGB or SG. The surgical risk, the differential impact of each procedure on body weight and other obesity-related diseases, presence of other medical and mental problems, patient's behavioral factors (e.g., postoperative compliance, active smoking), medications, and goals will be considered when the patient and local medical team make a shared decision about the most appropriate surgical procedure.
  Other Names: Metabolic Surgery; Roux-en-Y Gastric Bypass (RYGB); Sleeve Gastrectomy (SG)
  Arms: Bariatric Surgery
Drug: Semaglutide — Semaglutide will be initiated at a dose of 0.25 mg once weekly and will be increased during the dose-escalation period to reach a maintenance dose of up to 2.4 mg once weekly by week 16. If patients do not tolerate a dose during dose escalation, we will consider delaying dose escalation until next visit (for 4 weeks). Dosing for Semaglutide is the FDA-approved dosing schedule.
  The maintenance dose is 2.4 mg injected subcutaneously once-weekly. The protocol allows for dose reductions in case a participant does not tolerate the recommended target dose of 2.4 mg and may stay at the lower maintenance dose level (e.g., 1.7 mg once weekly), if needed.
  Other Names: Ozempic; Wegovy
  Arms: Semaglutide
Drug: Tirzepatide — Tirzepatide will be initiated at a dose of 2.5 mg once weekly and will be increased by 2.5 mg every week during the dose-escalation period to reach a maintenance dose of up to 15 mg once weekly by week 20. If patients do not tolerate a dose during dose escalation, we will consider delaying dose escalation until next visit (for 4 weeks). Dosing for Tirzepatide is the FDA-approved dosing schedule.
  The maintenance dose is 15 mg injected subcutaneously once-weekly. The protocol allows for dose reductions in case a participant does not tolerate the recommended target dose of 15 mg and may stay at the lower maintenance dose level (e.g., 10 mg once weekly), if needed.
  Other Names: Mounjaro; Zepbound
  Arms: Tirzepatide

SUMMARY:
The recent introduction of the new generation of anti-obesity medications (AOMs) will change the future of obesity treatment. These highly effective medications, such as high-dose semaglutide and tirzepatide, are hormone analogues that augment the incretin function and exert multiple physiological effects by activating glucagon-like peptide-1 (GLP-1) and/or glucose-dependent insulinotropic polypeptide (GIP) distributed in various organs. These medications provide an average of 15-22% weight reduction in one-year trials, which had not been seen in the past with medical therapy. While the literature suggests that bariatric surgery is superior to these new highly effective medications, there is no head-to-head comparison between the most common bariatric operations (Roux-en-Y gastric bypass [RYGB] and sleeve gastrectomy [SG]) with semaglutide (once weekly) and tirzepatide (once weekly). The goal of this Randomized Clinical Trial (RCT) is to compare these effective therapies in patients with severe obesity to provide the best evidence to inform clinical decisions in treating patients with obesity.

DETAILED DESCRIPTION:
This is a randomized, non-blinded, controlled efficacy/safety study with 3 parallel groups who will either receive bariatric surgery (RYGB or SG), semaglutide, or tirzepatide. The study has 2 phases: the first 12 months for the assessment of the primary endpoint ( mean percentage weight loss) and the second 12 months as the extension phase of the study to mimic the real-life setting. Findings at the end of each phase will be separately reported.

A randomized trial of 125 patients with a BMI of 35-65 kg/m2 who sought treatment for obesity at Cleveland Clinic will be performed. Patients who meet the ASMBS/IFSO 2022 guidelines for bariatric surgery will be invited for possible enrollment. Interested and eligible patients will be randomized to receive their already chosen bariatric surgery (RYGB or SG), tirzepatide. or semaglutide in 2:2:1 ratio.

The study is not intended to compare RYGB vs SG head-to-head. RYGB and SG constitute one group as a bariatric surgery group. The assignment of RYGB or SG is not based on a randomized design. Each patient and surgical team will make a shared decision about the most appropriate surgical procedure. The study is also not intended to compare semaglutide vs tirzepatide head-to-head.

In the second or extension phase of the study, participants are followed from month 12 to month 24, regardless of the treatment that they receive. In this phase, the study medications (semaglutide and tirzepatide) will not be provided by the study. The goal of this phase is to provide valuable insights into A) access to AOMs and the durability of effects in the real-life setting, B) cross-over from AOMs to bariatric surgery, and C) adjuvant pharmacotherapy after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

Entry into the study would require that the patient:

1. Is a candidate for general anesthesia
2. Is eligible for bariatric surgery (RYGB or SG) based on ASMBS/IFSO 2022 guidelines
3. Is ≥18 and ≤70 years old (both inclusive)
4. has a BMI ≥35 and ≤65 kg/m2 (both inclusive)
5. Patients with and without T2DM are eligible for the study. Patients with T2DM should have been on a stable dose of anti-diabetic medication (including insulin but not semaglutide or tirzepatide) for at least 3 months prior to entry, with HbA1c ≤12%.
6. No weight loss > 20 lbs. in 3 months before screening (self-reported)
7. Has the ability and willingness to participate in the study, provide informed consent, and agree to any of the arms involved in the study.
8. Is able to understand the options and to comply with the requirements of each arm.
9. Has a negative urine pregnancy test at randomization visit for women of childbearing potential.
10. Women of childbearing age must agree to use reliable method of contraception for 2 years.

Exclusion Criteria:

1. Significant cardiac or atherosclerotic disease (planned to undergo cardiac, coronary, carotid, or peripheral artery revascularization procedures in the next 12 months)
2. Severe uncompensated cardiopulmonary disease leading to American Society of Anesthesiologists Class IV or V
3. Classified as New York Heart Association Class IV
4. Left ventricular ejection fraction <25% at the time of screening (if already known)
5. Myocardial infarction, unstable angina, stroke, transient ischemic attack, heart surgery, coronary stent placement in the past 6 months
6. Prior bariatric surgery of any kind

   • Intragastric balloon that has been removed at least 6 months prior to the first study visit is allowed.
7. History of solid organ transplant
8. Type 1 diabetes or autoimmune diabetes
9. eGFR < 30 mL/min/1.73 m2 or being on dialysis
10. History of deep vein thrombosis, pulmonary embolism, or venous thromboembolism
11. On therapeutic dose of anticoagulants such as warfarin or direct oral anticoagulants (DOACs)
12. Decompensated cirrhosis characterized by presence of ascites, hepatic encephalopathy, portal hypertension, or esophageal varices.
13. History of severe anemia defined as hemoglobin less than 8 g/dL
14. Use of investigational therapy
15. Liver transaminase level or alkaline phosphatase >200 U/L
16. Significant alcohol use (average >2 drinks/day)
17. Presence of active malignancy (except non-melanoma skin cancer)
18. Life expectancy less than 3 years due to concomitant diseases
19. Major mental health, psychological disorders, or substance abuse disorders that in the opinion of the investigators could disqualify the patient from bariatric surgery
20. Any condition or major illness that, in the investigator's judgment, places the subject at undue risk by participating in the study
21. Unable to understand the risks, benefits and compliance requirements of study
22. Lack capacity to give informed consent
23. Plans to move outside the primary location of study (northeast Ohio) within the next 12 months
24. Pregnant, breast-feeding or the intention of becoming pregnant or not using adequate contraceptive measures
25. Hypothalamic obesity
26. Continuous treatment with semaglutide (once weekly) or tirzepatide (once weekly) <60 days before screening
27. History of semaglutide (once weekly) or tirzepatide (once weekly) use in the past for obesity with lack of clinical response
28. Chronic use of systemic steroids
29. Uncontrolled thyroid disease: thyroid stimulating hormone (TSH) > 6.0 mIU/L or < 0.1 mIU/L

    • Note: Patients receiving treatment for hypothyroidism can be included if their thyroid hormone replacement dose has been stable for at least 3 months.
30. Acute pancreatitis < 180 days before screening
31. History or presence of chronic pancreatitis
32. History of Crohn's disease
33. Known or suspected allergy to semaglutide, tirzepatide, excipients, or related products
34. A personal or family history of medullary thyroid carcinoma (MTC) or in patients with Multiple Endocrine Neoplasia syndrome type 2 (MEN 2)
35. Previous participation in this trial and got randomized to one of the study groups but did not proceed.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
The mean percentage weight loss | First 52 weeks of the study
  The mean percentage weight loss at 52 weeks for the following 2 comparisons:
  * Bariatric surgery (RYGB and SG) vs tirzepatide
  * Bariatric surgery (RYGB and SG) vs semaglutide

SECONDARY OUTCOMES:
Percentage of Participants Achieving Weight Loss Milestones (Body weight related end points) | First 52 weeks of the study
  Percentage of participants achieving ≥5%, ≥10%, ≥15%, ≥20%, ≥25%, ≥30%, and ≥35% weight loss from baseline
Absolute Change in Weight (Body weight related end points) | First 52 weeks of the study
  Mean absolute change in weight measured in kilograms from baseline to 52 weeks
Absolute Change in BMI (Body weight related end points) | First 52 weeks of the study
  Absolute change in BMI measured in kg/m^2 from baseline to 52 weeks
Excess Weight Loss Percentage (Body weight related end points) | First 52 weeks of the study
  Percentage of excess weight loss, calculated by dividing the difference between initial BMI and final BMI by the difference between initial BMI and a target BMI of 25
Change in Waist Circumference (Body weight related end points) | First 52 weeks of the study
  Change in waist circumferential measurement above the level of the iliac crests measured in centimeters from baseline to 52 weeks
Systolic blood pressure trends | First 52 weeks of the study
  Mean and change in systolic blood pressure measured in mmHg
Mean and change from baseline in lipid panel | First 52 weeks of the study
  Mean and change from baseline in total cholesterol, high-density lipoprotein (HDL), low-density lipoprotein (LDL), and triglycerides
Changes in glucose homeostasis markers in T2DM patients | First 52 weeks of the study
  Mean and change from baseline in blood glucose and HbA1c in patients with T2DM
Percentage of patients with T2DM meeting predefined HbA1c targets | First 52 weeks of the study
  Percentage of patients meeting different HbA1c targets, for example:
  * HbA1c <6.5% (without diabetes medications)
  * HbA1c <7% (irrespective of taking diabetes medications or not)
Changes in inflammatory marker, CRP | First 52 weeks of the study
  Mean and change from baseline in C-Reactive Protein (CRP) measured in mg/L
Changes in Lipoprotein(a) | First 52 weeks of the study
  Mean and change from baseline in Lipoprotein(a) measured in mg/dL
Change in cardiovascular and diabetes medications | First 52 weeks of the study
  Change in the number of cardiovascular and diabetes medications prescribed
Change from baseline in quality of life metrics | First 52 weeks of the study
  Change from baseline in score of The 36-Item Short Form Health Survey (SF-36) (physical and mental components). Each item is given a score ranging from 0-100. Lower scores indicating poor outcomes. Final score is an average of all the items that were answered. Unanswered questions are not included in the final average. Research coordinator completes the survey with the patient.
Change in body composition (via Seca mBCA 554 Bioimpedance Analysis) | First 52 weeks of the study
  Change in body composition (% fat mass and % fat-free mass) as measured by Seca mBCA 554 Bioimpedance Analysis to assess whether that weight loss is primarily caused by reduction in fat mass or not.
Mean change in liver fat content (via MRI-PDFF) | First 52 weeks of the study
  Mean change from baseline in liver fat content as assessed by MRI-PDFF measured as a percentage
Percentage of Participants Achieving ≥5%, ≥30%, ≥50% Absolute Reduction in Liver Fat Content (via MRI-PDFF) | First 52 weeks of the study
  Percentage of participants achieving at least 5%, 30%, or 50% relative reduction in liver fat content from baseline
Percentage of Participants Achieving MRI-PDFF Normalization (via MRI-PDFF) | First 52 weeks of the study
  Percentage of participants achieving MRI-PDFF normalization, defined as a liver fat content of <5%, at week 52

OTHER OUTCOMES:
Cardiac ejection fraction (via cardiac MRI) | First 52 weeks of the study
  Ejection fraction of the heart evaluated via cardiac MRI measured in percentage
Left ventricular mass (via cardiac MRI) | First 52 weeks of the study
  Left ventricular mass, evaluated via cardiac MRI measured in grams
Pericardial fat fraction (via cardiac MRI) | First 52 weeks of the study
  fat fraction of the pericardium via cardiac MRI measured in percentage
change in body weight (second phase of the study) | from week 52 to week 104 of the study
  Change in body weight in percentage during the extension phase of the trial mimicking what can happen in the real-life setting
Cross-overing to bariatric surgery (second phase of the study) | from week 52 to week 104 of the study
  Percentage of patients cross-over from nonsurgical arm to bariatric surgery
Anti-obesity medication after bariatric surgery (second phase of the study) | from week 52 to week 104 of the study
  Percentage of patients receiving anti-obesity medications after bariatric surgery
Change in body weight in patients receiving combination therapy (second phase of the study) | from week 52 to week 104 of the study
  Change in body weight in percentage during the extension phase of the trial in the patients who receive both bariatric surgery and anti-obesity medications
Safety end points | Throughout the study, 104 weeks
  Complications related to obesity, bariatric surgery, as well as adverse events of semaglutide and tirzepatide in the trial will be recorded and evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Aminian, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No